CLINICAL TRIAL: NCT03236298
Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: a RCT Comparing 125 mL/h Versus 250 mL/h Bolus Delivery Flow
Brief Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: Comparing 125 mL/h Versus 250 mL/h Bolus Delivery Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-02
Record Dates: First submitted 2017-07-12; First posted 2017-08-01 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Labor Pain
Keywords: Epidural; Labor analgesia; Programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIEB speed of infusion 250 ml/hr (Active Comparator): The programmed intermittent bolus of 10ml will be administered every 40 minutes, at a speed of 250 ml/hr by the CADD-Solis Ambulatory Infusion System.
  Interventions: Device: CADD-Solis Ambulatory Infusion System
- PIEB speed of infusion 125 ml/hr (Active Comparator): The programmed intermittent bolus of 10ml will be administered every 40 minutes, at a speed of 125 ml/hr by the CADD-Solis Ambulatory Infusion System.
  Interventions: Device: CADD-Solis Ambulatory Infusion System

INTERVENTIONS:
Device: CADD-Solis Ambulatory Infusion System — The CADD-Solis pump will administer programmed intermittent boluses of 0.0625% Bupivacaine plus fentanyl 2mcg/ml.

SUMMARY:
At Mount Sinai Hospital, epidural analgesia for labor pain is delivered by programmed intermittent epidural bolus (PIEB), in combination with pushes of medication activated by the patient, a technique called patient controlled epidural analgesia (PCEA). Studies have shown that delivering analgesia in this manner can prolong the duration of analgesia, diminish motor block, lower the incidence of breakthrough pain, improve maternal satisfaction and decrease local anesthetic consumption comparing to a conventional continuous infusion. The use of this PIEB technique in routine practice has reduced the total consumption of local anesthetic and the percentage of patients requesting additional boluses (PCEA or manual rescues).

However, at the same time, sensory blocks above those targeted for labor pain relief have been reported in our institution, suggesting that the spread of the freezing medication is wider than necessary. Based on the information already available in the literature, the investigators will conduct this study to determine the best regimen of PIEB achievable with a slower delivery speed.

The hypothesis of this study is that PIEB boluses with 125 mL/h will decrease by 50% the incidence of women presenting sensory block to ice equal or higher than T6 as compared to a delivery rate of 250 mL/h.

DETAILED DESCRIPTION:
PIEB is a novel technique, which provides better analgesia and less motor block; however, the ideal regimen has not been established. To optimize the PIEB regimen, the investigators have conducted several clinical trials using bupivacaine with fentanyl. Although PIEB provides the excellent analgesia to laboring parturients, studies completed by the instigators have shown that the incidence of sensory block to ice ≥T6 was 66%. For labor analgesia during the first stage of labor, effective sensory block requires T10 to L1; therefore, a sensory block ≥T6 seems unnecessarily high, and the investigators seek to confine epidural spread within a proper range.

Our previous studies showed that the effective volume 90% using 0.0625% bupivacaine was 10.7 mL, and incidence of epidural blockade ≥T6 was similar even using a 5-mL bolus with 0.125% bupivacaine. The investigators concluded that it is not possible to reduce volume of the PIEB, or use a higher concentration of local anesthetic without compromising the quality of analgesia. There is some evidence in the literature that supports the idea that higher injection pressures result in a wider spread of local anesthetic administered into the epidural space, therefore a slower epidural delivery flow rate may result in less spread.

ELIGIBILITY:
Inclusion Criteria:

* ASA II or III
* Term pregnancy (gestational age ≥ 37 weeks)
* Nulliparous
* Singleton pregnancy with vertex presentation
* Active labour defined as occurring regular uterine contractions at least every 5 minutes with progressive cervical dilatation
* Verbal Numerical Rating Score (VNRS) greater than 5 at requiring epidural analgesia (VNRS 0-10)
* Cervical dilation between 2 and 5 cm

Exclusion Criteria:

* Any contraindication to epidural analgesia
* Accidental dural puncture
* Drug allergy to lidocaine, bupivacaine or fentanyl
* Use of pharmacological analgesics within the last 4 hours
* Patient refusal to participate in the trial

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Sensory block level to ice equal to or higher than T6 within the study period (6 hours) | 6 hours
  Sensory block to ice will be assessed bilaterally at the mid-clavicular line, and the level of block will be the level at which the patient still does not feel normal cold sensation as compared to a control site (lateral upper arm, frontal part of head or cheek). T6 is defined as the level of the xyphoid process.

SECONDARY OUTCOMES:
Sensory block level to ice | 6 hours
  Sensory block to ice will be assessed bilaterally at the mid-clavicular line hourly (for up to 6 hours), and the level of block will be the level at which the patient still does not feel normal cold sensation as compared to a control site (lateral upper arm, frontal part of head or cheek).
Sensory block level to pin prick | 6 hours
  Sensory block to pin prick will be assessed bilaterally at the mid-clavicular line hourly (for up to 6 hours), and the level of block will be the level at which the patient initial begins to feel normal sharp sensation compared to a control site (lateral upper arm, frontal part of head or cheek).
Motor block level assessed using Bromage score | 6 hours
  Motor block will be assessed hourly with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle.
Pain score | 6 hours
  Pain score measured hourly (for up to 6 hours) using VNRS (0-10)
Total number of PCEA demands | 6 hours
  The number of times a patient presses the button to request additional analgesia.
Total number of rescue boluses administered | 6 hours
  The number of actual boluses administered by the patient, nurse or physician (for up to 6 hours).
Total amount of local anesthetic (ml) | 6 hours
  The total amount of local anesthetic consumption over the study period (by programmed intermittent bolus and any rescue boluses, for up to 6 hours).
Maternal satisfaction rating | 6 hours
  Maternal satisfaction rating using VNRS (0-10), 0=not at all satisfied, 10=most satisfied Rating at the end of the 6 hour study period.
Hypotension | 6 hours
  A decrease in systolic blood pressure greater than 20% from baseline (defined as an average of 3 readings prior to epidural), during the 6 hour study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazda Y, Arzola C, Downey K, Ye XY, Carvalho JCA. Programmed intermittent epidural bolus for labour analgesia: a randomized controlled trial comparing bolus delivery speeds of 125 mL.hr-1 versus 250 mL.hr-1. Can J Anaesth. 2022 Jan;69(1):86-96. doi: 10.1007/s12630-021-02132-w. Epub 2021 Nov 1. PMID 34725792